CLINICAL TRIAL: NCT04281719
Title: M-Health for Teen Substance Abuse and Mental Illness: Component III
Brief Title: M-Health for Teen Substance Abuse and Mental Illness Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unanticipated technical issues and COVID-19 related-disruptions precluded enrollment of participants before the end of the award period.
Sponsor: Indiana University (Other)
Collaborators: Health Information Technology Solutions (HITS) LLC (Unknown)
Responsible Party: Principal Investigator, Zachary W. Adams, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1908720822
Record Dates: First submitted 2020-01-31; First posted 2020-02-24 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Substance Use Disorders; Post Traumatic Stress Disorder; Adolescent Behavior; Mental Health Disorder
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic; Adolescent Behavior; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile App (Experimental): Youth will be assigned to interact with a novel mobile application during a course of outpatient psychotherapy for substance use disorder(s) and co-occurring mental health disorder(s).
  Interventions: Other: Mobile Application (working name: Bright Path)

INTERVENTIONS:
Other: Mobile Application (working name: Bright Path) — The Bright Path web-based mobile application is designed to target co-occurring problems, enhance patient treatment engagement, and contribute to lasting improvements in teens' mental health. The central hypothesis is that developmentally tailored mobile applications that incorporate evidence-based treatment principles can facilitate increased patient engagement in and between sessions, thus, improving the efficiency, efficacy, and reach of treatments for this highly vulnerable population.

SUMMARY:
The study is exploring the ease and ability to integrate a mobile application in outpatient behavioral health treatment. There are two major aims to the study: 1) Determine feasibility and acceptability of integrating a mobile app into behavioral health treatment for adolescents with co-occurring substance use and mental health disorders, and 2) identify initial signal of effect on engagement and/or treatment outcomes among youth who use the mobile app.

DETAILED DESCRIPTION:
The purpose of the trial will be to demonstrate the feasibility of the proposed methodology (rate of recruitment, retention at 4-month follow-up, study procedures) as well as estimates of effect on key variables (patient engagement, patient symptoms, use of e-tools, treatment efficiency) in preparation for future studies in this line evaluating the utility of the mobile app.

ELIGIBILITY:
Inclusion Criteria for Adolescents:

* Aged 14-17 years
* Current substance use disorder (SUD)
* Co-occurring mental health disorder
* Treatment-seeking
* English-speaking (Only English documents will be used throughout the course of this research study)

Exclusion Criteria for Adolescents:

* Younger than 14 or older than 17
* Endorsement of active suicidal or homicidal ideation
* Active mania or psychosis
* Significant cognitive disability, developmental delays, or pervasive developmental disability
* No history of outpatient psychotherapy.

Inclusion Criteria for Providers

* Clinician delivering outpatient dual diagnosis treatment (i.e., for co-occurring SUDs and mental health disorders)
* Therapist with at least a Master's degree in a counseling related field

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients retained in study protocol | 4 months post-baseline
  Retention of >75% of adolescents through assessments measured by study participant enrollment records. The retention rate will be measured by the number of sessions attended.
Provider satisfaction assessed by Treatment Evaluation Inventory-Short Form (TEI-SF) | 4 months post-baseline
  Providers express high satisfaction with e-tools per published norms on the TEI-SF. The Treatment Evaluation Inventory Short Form (TEI-SF) is a 9-item questionnaire that is rated on a 5-point scale. Scores range from 9 to 45 for each treatment with higher scores indicating greater acceptability of the model.
Adolescent satisfaction assessed by the Client Satisfaction Questionnaire (CSQ) | 4 months post-baseline
  Adolescents express high satisfaction with e-tools per published norms. The Client Satisfaction Questionnaire-8, an 8 question survey with ratings from 1 to 4 is used. Scores can range from 8 to 32 with higher scores indicating greater satisfaction.
Patient Engagement assessed by the Child Improvement Rating Scale (CIRS) | 4 months post-baseline
  Provider-rated youth engagement in treatment process.This will be assessed by the Child Involvement Rating Scale (CIRS) which is a 6 item questionnaire with each item being rated on a 6 item scale ranging from 0 to 5. The questionnaire contains 4 items assessing positive involvement and 2 items assessing negative involvement. The positive items are scored according to the selected scale value while the negative involvement items are reverse scored. Higher scores correspond to greater perceived patient involvement.

SECONDARY OUTCOMES:
Substance Use Disorder (SUD) Symptoms measured by CRAFFT | 4 months post-baseline
  Providers record a decrease in SUD symptoms for patients participating in the study and treatment. The CRAFFT, a 6-item questionnaire in which every "yes" scores 1 point is used to measure substance abuse and dependence. A score of 2 or higher indicates a positive screening.
Substance Use Disorder (SUD) Symptoms assessed by the Drug Abuse Screening Test for Adolescents (DAST-20-A) | 4 months post-baseline
  Providers record a decrease in SUD symptoms for patients participating in the study and treatment. The Drug Abuse Screening Test-20 Adolescent Version (DAST-20-A) is a 20-item self-report questionnaire. Higher scores indicate a greater severity in substance use and can be broken down into the following ranges: 0 (n/a), 1-5 (low), 6-10 (intermediate, likely meets DSM criteria), 11-15 (substantial), 16-20 (severe).
Post-Traumatic Stress Disorder (PTSD) Symptoms (If applicable) | 4 months post-baseline
  Providers record a decrease in PTSD symptoms for patients participating in the study and treatment. The PTSD Symptom Scale for DSM-5 (CPSS-5) is used for evaluation. The CPSS-5 is a 20-item symptom checklist in which symptom severity can be rated from 0 to 4. Higher scores indicate greater symptom severity and can be broken down into the following ranges: 0-10 (minimal), 11-20 (mild), 21-40 (moderate), 41-60 (severe), 61-80 (very severe)
Therapeutic alliance as measured by the Therapeutic Alliance Scale for Children-Revised (TASC-R) | 4 months post-baseline
  Providers record high therapeutic alliance per published norms. The TASC-R includes 12 items rated on a Likert scale from 1 (not true) to 4 (very much true), with item scores summed for a total, where higher scores correspond to higher therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary W Adams, PhD, Principal Investigator — Indiana University School of Medicine